CLINICAL TRIAL: NCT06531213
Title: Effects of Visual Perception Intervention Programme on Fine Motor and Visual Perception in Children With Down Syndrome
Brief Title: Visual Perception Intervention Programmes Impact on Down Syndrome Affiliate Children's Fine Motor and Visual Perception.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07101
Record Dates: First submitted 2024-06-11; First posted 2024-07-31 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Down Syndrome
Keywords: down syndrome; visual motor skills; Fine motor skills; postural instability
MeSH Terms: conditions — Down Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: it will be randomized control trail in which nonprobability convenient sampling will be used .two groups 5 to 9 age will be formed in which participants will randomly divided.
  Experimental Group: Baseline rehabilitation, Visual Perception Interventions. Control Group: Home-based activities, Baseline Rehabilitation (strengthening exercise, achieving missing milestones).
Who Masked: Participant
Masking Description: single participant will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Visual Perception Activities and usual care group
  Interventions: Other: experimental
- Group B (Experimental): Usual Care group (control)
  Interventions: Other: controlled

INTERVENTIONS:
Other: experimental — Experimental Group: Baseline rehabilitation, Visual Perception Interventions. Home base activities, Baseline Rehabilitation (Strengthing exercise, achieving missing milestones).
  Visual Perception Interventions
  • Puzzle:Give step-by-step • printable activities • Sudoku. SET, Search Word, Spot it, what is missing, Tic Tac Toe, I Spy
  Arms: Group A
Other: controlled — Controlled: Baseline rehabilitation. Home-based activities, Baseline Rehabilitation (strengthening exercise, achieving missing milestones).3. Activities Play Dough ( Manipulation) Draw on sketch Cup stacking.
  Other Names: usual control group
  Arms: Group B

SUMMARY:
A second copy of chromosome 21 results in Trisomy 21, a genetic disorder commonly referred to as Down syndrome. In addition to physical traits like low muscular tone, upward-slanting eyes, and a flat facial profile, this extra genetic material causes intellectual and developmental difficulties. Even though people with Down syndrome may experience a range of health problems, they can lead happy, fulfilling lives if they receive the right support and care. Individual differences in the illness's severity are significant.

There will be a randomized control trial. People with Down syndrome who are five to nine years old will be screened for this study. Adults with Down syndrome and severe ID will not be eligible to participate in this study. Participants will be selected using

DETAILED DESCRIPTION:
Conventional physical therapy will be administered to the participants in both groups. Visual perception interventions will be administered to the intervention group, and then standard treatment will follow. For six weeks, there will be three 45-minute treatment sessions per week. Using outcome measure instruments, data will be gathered twice: once at the beginning of the study and again at the end of the six-week course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between 6-9 years.
* IQ level mild to moderate (below 40)

Exclusion Criteria:

* Heart,
* GIT problems,
* respiratory problems
* and hearing loss.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Berry Visual Motor Integration | 8weeks
  The berry VMI is designed to assess a person's ability to integrate visual and motor skills so that the proper treatment can be provided
Bruininks oseretsky test | 8weeks
  BOT-2 measures fine and gross motor proficiency, with subtests that focus on stability, mobility, strength, coordination, and object manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Zohaib Saddiquee, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahin S, Kose B, Aran OT, Bahadir Agce Z, Kayihan H. The Effects of Virtual Reality on Motor Functions and Daily Life Activities in Unilateral Spastic Cerebral Palsy: A Single-Blind Randomized Controlled Trial. Games Health J. 2020 Feb;9(1):45-52. doi: 10.1089/g4h.2019.0020. Epub 2019 Jul 23. PMID 31335174